CLINICAL TRIAL: NCT05499572
Title: Usability of Levodopa Cyclops™ Compared to INBRIJA® During an Off Episode in Parkinson's Disease Patients
Brief Title: Usability of Levodopa Cyclops™ vs INBRIJA® in Parkinson's Patients
Acronym: DPI-6
Status: Completed | Type: Observational
Sponsor: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL82043.099.22
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Usability
Keywords: Parkinson

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inbrija followed by Cyclops: During an off episode, patients will demonstrate both inhaler user maneuvers. The researcher will observe whether the steps are followed correctly. The handling time will be recorded as well. To see whether the patients prefer a certain inhaler and to see where this preference comes from, they need to fill in a questionnaire. The questionnaire will be filled in during or directly after the off episode. Dummy inhalers are used, so patients will only inhale air (no medication).
  Interventions: Device: Inhalation maneuver with placebo Inbrija and placebo Cyclops
- Cyclops followed by Inbrija: During an off episode, patients will demonstrate both inhaler user maneuvers. The researcher will observe whether the steps are followed correctly. The handling time will be recorded as well. To see whether the patients prefer a certain inhaler and to see where this preference comes from, they need to fill in a questionnaire. The questionnaire will be filled in during or directly after the off episode. Dummy inhalers are used, so patients will only inhale air (no medication).
  Interventions: Device: Inhalation maneuver with placebo Inbrija and placebo Cyclops

INTERVENTIONS:
Device: Inhalation maneuver with placebo Inbrija and placebo Cyclops — Patients perform the inhalation maneuvers with placebo inhalers (Inbrija and Cyclops) during a Parkinson's off episode.

SUMMARY:
Currently there is one Levodopa inhaler on the market, the INBRIJA® inhaler. When looking at the user instructions for the INBRIJA®, multiple steps are necessary including preparing and cleaning the inhaler. The Levodopa Cyclops™ inhaler also requires steps to be ready-for-use, however there are less steps required to reach this 'ready-for-use' state. This is mainly because the medicine (Levodopa) is already prefilled in the inhaler. Moreover, the Levodopa Cyclops™ is a single-use inhaler and cleaning steps are not necessary. Since both inhalers should be used during off episodes, there might be a preference for one inhaler over the other due to the instructions. An off episode might impair the ability and length to successfully operate an inhaler due to mental or mobility issues. This study investigates if Parkinson patients have a preference for one of the inhalers based on handling steps, ease-of-use, understandability.

DETAILED DESCRIPTION:
Sixteen Parkinson's patients, who are ≥ 18 years of age, regularly suffering from predictable off episodes, able to understand the inhaler user instructions (no cognitive dysfunction) and who did not previously participate in the Parkinson DPI-1,2,3,4 or 5 study or in a study using INBRIJA®.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease by a neurologist;
* At least 18 years of age;
* Regularly suffering from predictable off episodes despite medication;
* Recognizable off episodes for themselves and others;
* Signed informed consent

Exclusion Criteria:

* Not able to understand an inhalation instruction of either the Levodopa Cyclops™ or the INBRIJA® (within a maximum of 20 minutes of explanation per inhaler);
* Cognitive dysfunction, which precludes good understanding of instructions and/or informed consent;
* Previously participated in the Parkinson DPI-1, DPI-2, DPI-3, DPI-4 or DPI-5 study (prior knowledge of the inhalation maneuver of the Levodopa Cyclops™)
* Having experience with using the INBRIJA® inhaler.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Correct performance of inhalation maneuvers | 15 minutes for performing the inhalation maneuvers with both the placebo inhalers (Inbrija and Cyclops) during a Parkinson's off episode
  The main study parameter is to investigate whether Parkinson's patients perform the correct steps in accordance with the instruction card of respectively the Levodopa Cyclops™ or INBRIJA® inhaler after the primary inhalation instructions.

SECONDARY OUTCOMES:
Inhaler preference of Parkinson patients | 10 minutes for filling in the questionnaire during or directly after a Parkinson's off episode
  The secondary study parameter is to investigate whether the Parkinson's patients prefer the Levodopa Cyclops™ or the INBRIJA® inhaler by keeping track of the total handling time and by letting the patients fill in a questionnaire keeping track of their experiences regarding the ease-of-use, convenience and preference of the different steps of the inhaler user maneuver

CONTACTS AND LOCATIONS:
Locations (1):
- Martini Ziekenhuis, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No